CLINICAL TRIAL: NCT06187545
Title: Clinical Performance of a Minimum Viable Prototype for Automated Closed-Loop Administration of Propofol for Deep Sedation in Patients on Invasive Mechanical Ventilation in Critically Ill Patient Units: a Pilot Randomized Clinical Trial
Brief Title: Clinical Performance of the Automated Closed-loop Minimum Viable Prototype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1219/21
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Deep Sedation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 5-hour period in which patients will continue to be routinely sedated in the critical care unit
  Interventions: Device: Usual care
- Experimental group (Experimental): 5-hour period in which patients will be sedated through the closed-loop system
  Interventions: Device: Minimum viable prototype

INTERVENTIONS:
Device: Minimum viable prototype — Deep sedation in critical ill patients using minimum viable prototype
  Arms: Experimental group
Device: Usual care — Deep sedation without minimum viable prototype
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate a minimum viable prototype for automated closed-loop administration of propofol in deep sedated patients under invasive mechanical ventilation in the ICU. The main question it aims to answer is:

• whether the minimum viable prototype for automated closed-loop administration of propofol is effective in keeping patients in deep sedation using the lowest possible dose of propofol Participants will undergo deep sedation using the minimum viable prototype for automated closed-loop propofol administration.

The usual practice of sedation will be compared with the practice of sedating with the minimum viable prototype to see if the infusion rate of propofol is decreased

DETAILED DESCRIPTION:
The design of the study will consist of each patient being exposed to both forms of administration (matched pair study) during a 12-hour day (8:00 a.m. to 8:00 p.m.) in a randomized manner. Specifically, a patient will be given propofol infusion in open-loop mode in the first 5 hours (8:00 a.m. to 1:00 p.m.) and the next 5 hours in closed-loop mode (3:00 p.m. to 8:00 p.m.) with a wash-out period of 2 hours. The order will be randomly determined for each patient. This design will allow the use of the prototype to be evaluated under highly controlled conditions by a trained operator dedicated exclusively to this function.

ELIGIBILITY:
Inclusion Criteria:

* Indication of deep sedation for more than 48 hours

Exclusion Criteria:

* Dementia
* Cranial surgery
* Hypoxic-ischemic encephalopathy
* Chronic liver damage Child C
* History of substance and drug abuse that can alter EEG recordings or the metabolization of drugs (antipsychotics, cocaine, benzodiazepines, opioids)
* Pregnant women
* allergic to propofol
* EEG sensor of the BIS® Covidien cannot be installed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Infusion rate of propofol | Fifth hour
  mg/kg/h

SECONDARY OUTCOMES:
Sedation level | Fifth hour
  Scale SAS (Sedation-Agitation Scale, Score 1-7) (1-2 deeply sedated, 3-4 sedated or calm, 5-6 agitated, and 7 dangerously agitated)
Total dose of propofol | Five hours
  mg
BIS level | Five hours
  BIS index (bispectral index, values from 0-100, 0 is the minimum, which indicates isoelectric electroencephalographic activity and 100 is the maximun, which indicates awake electroencephalographic activity)
Suppression rate | Five hours
  Percentage
Norepinephrine infusion rate | fifth hour
  mcg/kg/min

CONTACTS AND LOCATIONS:
Locations (3):
- Chile (3):
  - Hospital Base San José Osorno, Osorno, Los Lagos Region
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: No